CLINICAL TRIAL: NCT06066424
Title: Phase 1 Dose Escalation and Expansion Study of TROP2 CAR Engineered IL15-transduced Cord Blood-derived NK Cells in Patients With Advanced Solid Tumors (TROPIKANA)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Bellicum Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-0161; NCI-2023-08351 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2023-09-27; First posted 2023-10-04 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Solid Tumors
MeSH Terms: interventions — fludarabine phosphate; fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose Escalation (Experimental): Participants who are enrolled in Dose Escalation, Participants will be assigned to a dose level of TROP2- CAR-NK cells based on when you join this study. Up to 5 dose levels of TROP2-CARNK cells will be tested. At least 3 participants will be enrolled at each dose level.
  The first group of participants will receive the lowest dose level. Each new group will receive a higher dose than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of TROP2-CAR-NK cells is found.
  Participants who are enrolled in the Dose Expansion, Participants will receive TROP2-CAR-NK cells at the recommended dose that was found in the Dose Escalation.
  Interventions: Drug: Rimiducid; Drug: TROP2-CAR-NK Cells; Drug: Fludarabine phosphate; Drug: Cyclophosphamide
- Dose Expansion Cohort 1 (Experimental): Participants who are enrolled in Dose Escalation, Participants will be assigned to a dose level of TROP2- CAR-NK cells based on when you join this study. Up to 5 dose levels of TROP2-CARNK cells will be tested. At least 3 participants will be enrolled at each dose level.
  The first group of participants will receive the lowest dose level. Each new group will receive a higher dose than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of TROP2-CAR-NK cells is found.
  Participants who are enrolled in the Dose Expansion, Participants will receive TROP2-CAR-NK cells at the recommended dose that was found in the Dose Escalation.
  Interventions: Drug: Rimiducid; Drug: TROP2-CAR-NK Cells; Drug: Fludarabine phosphate; Drug: Cyclophosphamide
- Dose Expansion Cohort 2 (Experimental): Participants who are enrolled in Dose Escalation, Participants will be assigned to a dose level of TROP2- CAR-NK cells based on when you join this study. Up to 5 dose levels of TROP2-CARNK cells will be tested. At least 3 participants will be enrolled at each dose level.
  The first group of participants will receive the lowest dose level. Each new group will receive a higher dose than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of TROP2-CAR-NK cells is found.
  Participants who are enrolled in the Dose Expansion, Participants will receive TROP2-CAR-NK cells at the recommended dose that was found in the Dose Escalation.
  Interventions: Drug: Rimiducid; Drug: TROP2-CAR-NK Cells; Drug: Fludarabine phosphate; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Rimiducid — Given by (IV) vein
Drug: TROP2-CAR-NK Cells — Given by (IV) vein
Drug: Fludarabine phosphate — Given by (IV) vein
  Other Names: Fludarabine; Fludara®
Drug: Cyclophosphamide — Given by (IV) vein
  Other Names: Cytoxan®; Neosar®

SUMMARY:
To find the recommended dose of TROP2- CAR-NK cells that can be given to participants with advanced forms of solid tumors.

DETAILED DESCRIPTION:
Primary Objective:

1. To determine the safety, tolerability, optimal cell dose (OCD), maximum tolerated dose (MTD), and recommended Phase 2 dose (RP2D) of TROP2-CAR-NK cells in participants with solid tumors with high TROP2 expression.

Secondary Objectives:

1. To determine the antitumor activity of TROP2-CAR-NK cells in participants with high TROP2-expressing NSCLC and high TROP2-expressing HER2-negative/low breast

   cancer. Although the clinical benefit of TROP2-CAR-NK cells has not yet been established, the intent of offering this treatment is to provide a possible therapeutic benefit and thus, the participant will be carefully monitored for tumor response and symptom relief in addition to safety and tolerability.
2. To quantify the persistence of infused allogeneic donor TROP2-CAR-NK cells in the peripheral blood of the recipient.
3. To evaluate tissue and blood-based biomarkers associated with response and resistance to TROP2-CAR-NK cell infusion.

Exploratory Objectives:

1. To profile and assess dynamic changes in the tumor microenvironment.
2. To evaluate longitudinal changes in circulating tumor DNA (ctDNA).

ELIGIBILITY:
Inclusion Criteria:

Patients must meet the following criteria for study entry:

1. Participants must be 18 years or older.
2. Participants must be willing and able to provide informed consent.
3. In the dose escalation, participants must have histologically documented locally advanced, unresectable, or metastatic solid tumor that has relapsed or progressed following local standard treatments that are known to prolong survival, or for which no standard treatment is available, or refused such therapy.
4. In dose expansion Cohort 1, patients must have histologically documented locally advanced, unresectable, or metastatic NSCLC. Participants should have received at least two prior lines of therapy in the advanced setting. Participants with metastatic PD-L1-positive disease will be expected to have prior immunotherapy unless contraindicated. Participants with actionable alterations (e.g., EGFR, ALK, BRAF V600E, RET, ROS1, MET, NTRK) should have received prior FDA-approved targeted therapy.
5. In dose expansion Cohort 2, patients must have histology documented locally advanced or metastatic HER2-negative/HER2-low breast cancer (IHC 0, IHC 1, or IHC 2+/ in situ hybridization negative) breast cancer. Participants should have received at least one prior line of therapy in the advanced setting. Participants with metastatic TNBC that is PD-L1 positive will be expected to have prior immunotherapy unless contraindicated. Participants with HR-positive disease will be expected to have received a prior cyclin- dependent kinase 4/6 inhibitor in the metastatic or adjuvant setting.
6. Participant tumors must demonstrate TROP2 expression of 2+ or 3+ as determined by IHC test at the MDACC Clinical Laboratory Improvements (CLIA) Laboratories (Clinical Lab or Clinical Translational Unit; Appendix 8).
7. Participants must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 (Appendix 3).
8. Life expectancy ≥3 months.
9. A female participant is eligible to participate if at least one of the following conditions applies:

   1. Not a woman of childbearing potential (WOCBP) as defined in Appendix 2 OR
   2. A WOCBP who agrees to follow the contraceptive guidelines in Appendix 2 during the study treatment period and for 6 months post TROP2-CAR-NK cell infusion.

   Female participants who become pregnant or suspect pregnancy must immediately notify their doctor. Females participants who become pregnant will be taken off study.
10. Male participants must agree to follow the contraceptive guidelines in Appendix 2 during the study treatment period and for 6 months post TROP2-CAR-NK cell infusion. Male participants who father a child or suspect that they have fathered a child must immediately notify their doctor.
11. WOCBP must have a negative urine pregnancy test within 72 hours prior to the start of lymphodepleting chemotherapy. If a WOCBP has a urine pregnancy test that cannot be confirmed as negative, a serum (beta-human chorionic gonadotropin [β-hCG]) pregnancy test will be required.
12. Participants must have measurable disease per the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 (Appendix 3).
13. Participants must have adequate organ function as defined below within 10 days prior to the start of lymphodepleting chemotherapy:

    Table 1. Adequate Organ Function Laboratory Values Systemic Function Test Laboratory Value Hematologic ANC ≥1500/µL Platelets ≥100,000/µL Hemoglobin ≥9.0 g/dLa Renal Creatinine OR CrCl by Cockcroft-Gault formula ≤1.5 × ULNb

    ≥45 mL/min for patients with creatinine >1.5 × ULNb Hepatic Total bilirubin ≤1.5 × ULN OR direct bilirubin ≤ ULN for patients with total bilirubin levels >1.5 × ULN AST and ALT ≤2.5 × ULN (≤5 × ULN for patients with liver metastases) Coagulation PT/INR aPTT ≤1.5 × ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants

    ALT=alanine aminotransferase; ANC=absolute neutrophil count; aPTT=activated partial thromboplastin time; AST=aspartate aminotransferase; CrCl=creatinine clearance; INR=international normalized ratio; PT=prothrombin time; ULN=upper limit of normal.
    1. Criteria must be met without erythropoietin dependency and without packed red blood cell transfusion within last 2 weeks of the screening test. Participants may be on a stable dose of erythropoietin (≥ approximately 3 months).
    2. Serum creatinine and CrCl should be interpreted and calculated per institutional standard.
14. Left ventricular ejection fraction >50%.
15. Adequate respiratory reserve defined as dyspnea Grade 0 or 1 and saturated oxygen >92% in room air.
16. Prior treatment with TROP2-targeted therapy will be allowed.
17. Willing to undergo mandatory blood collections and biopsies as required by the study.
18. Willing to sign consent for long-term follow-up on protocol PA17-0483.
19. Willing to stay within a 2-hour drive (approximately 100-mile radius) of the study site during the first 2 weeks after the TROP2-NK cell infusion.

Exclusion Criteria

Participants who meet any of the following criteria will not be eligible:

1. Pregnant, breastfeeding, or expecting to conceive within the projected duration of the study, starting with the screening visit through 6 months post TROP2-CAR-NK cell infusion.
2. Has received systemic anticancer therapy within 2 weeks or 5 half-lives, whichever is shorter, prior to the start of lymphodepleting chemotherapy. For participants treated with monoclonal antibodies, at least 3 weeks must have elapsed prior to the start of lymphodepleting chemotherapy. Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 3 weeks after the last dose of the previous investigational agent.
3. Participants must have recovered from all AEs due to previous therapies to ≤ Grade 1 or baseline. Participants with ≤ Grade 2 neuropathy, alopecia, or other non-relevant AEs may be deemed eligible at the discretion of the principal investigator (PI)/co-PIs. If a participant received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to the start of lymphodepleting chemotherapy.
4. Has received prior radiotherapy within 2 weeks of the start of lymphodepleting chemotherapy. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.
5. Has received a live vaccine within 6 weeks prior to TROP2-CAR-NK infusion and for at least 24 months post infusion. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin, and typhoid vaccine. Seasonal influenza and COVID- 19 vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist®) are live attenuated vaccines and are not allowed.
6. Prior CAR T or NK cell or other genetically modified T or NK cell therapy.
7. Has diagnosis of immunodeficiency or receiving chronic systemic steroid therapy (in doses exceeding 10 mg daily of prednisone equivalent).
8. History of a second malignancy, unless potentially curative treatment has been completed with no evidence of malignancy for 2 years. The time requirement does not apply to patients who underwent successful definitive resection of basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, in situ cervical cancer, or other in situ cancers.
9. Known active CNS metastases and/or carcinomatous meningitis. Patients with previously treated brain metastases may participate if they completed radiation therapy, are clinically stable, and without requirement of steroid treatment for at least 2 weeks prior to study enrollment.
10. Active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is allowed.
11. History of interstitial lung disease (ILD) that required steroids or has current pneumonitis/ILD.
12. Active infection requiring systemic therapy.
13. Known human immunodeficiency virus (HIV) infection.
14. Known active or chronic hepatitis B or hepatitis C virus infection.
15. Known history of active tuberculosis (Mycobacterium Tuberculosis).
16. History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the patient to participate, in the opinion of the treating investigator.
17. Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study.
18. Has had an allogenic tissue/solid organ transplant.
19. Clinically significant cardiovascular disease within 12 months prior to the start of lymphodepleting chemotherapy, including New York Heart Association Class III or IV congestive heart failure, unstable angina, myocardial infarction, cerebrovascular event, or cardiac arrhythmia associated with hemodynamic instability. NOTE: medically controlled arrhythmia would be permitted.
20. Prolongation of corrected QT interval using Fridericia's formula to >480 milliseconds.
21. Participants with bleeding or thrombotic disorders or at risk for severe hemorrhage. Participants with known deep vein thrombosis/pulmonary embolism who are on appropriate anti-coagulation treatment are eligible.
22. Participants with history of ≥ Grade 3 stomatitis or mucositis with prior therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-10-24 (Actual); Primary Completion 2038-04-30 (Estimated); Study Completion 2040-04-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0 | through study completion; an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ecaterina Dumbrava, M D, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org